CLINICAL TRIAL: NCT05821764
Title: Investigation of the Passage of Antiviral Antibodies From Mother to Child
Acronym: TransAc
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A01800-43
Record Dates: First submitted 2023-04-07; First posted 2023-04-20 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Pregnant Woman; Adult Patient
Keywords: Transfer; Placenta; Antibody; Virus
MeSH Terms: conditions — Virus Diseases | interventions — Blood Specimen Collection; Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Maternal blood (10ml) and cord blood (10ml)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The cohort for the TransAc study: Pregnant women followed for their pregnancy in the 3 Gynecology-Obstetrics department participating in the study
  Interventions: Other: Blood sample and data collection

INTERVENTIONS:
Other: Blood sample and data collection — Solicitation of parturients during a prenatal visit between 22 and 41 weeks of gestation or during their hospitalization in a high-risk pregnancy sector and at the latest on the day of their delivery.
  Blood sample :
  * Maternal sample within 72 hours before or after delivery during a care-based venipuncture (additional 10 mL sample) ;
  * The cord blood sample (10 mL) immediately after delivery.
  Data collection :
  * A data collection sheet for the attention of the investigator (doctor or midwife) ;
  * Additional data relating to the history of vaccination and infection completed by the patients included during their stay in the maternity ward and before their discharge from the hospital (Delay between 0 and 6 days after inclusion).

SUMMARY:
Infections remain a major cause of neonatal morbidity and mortality worldwide. At birth, multiple microorganisms, to which they are particularly vulnerable given the immaturity and naïve nature of their immune system, may infect newborns. Passive immunity by transplacental transfer of maternal antibodies is therefore of major importance in the first weeks and months of life before their own vaccination or until this period of immunological vulnerability has passed. Some factors are known to affect transplacental passage of antibodies but these have generally been studied in small series and many other parameters have not yet been investigated. The transmission rate of antibodies, particularly neutralizing antibodies, remains little explored, as well as the difference in transfer between antibodies induced by vaccination and those induced by natural infection, or the influence of maternal factors such as multiple pregnancy, other infections and treatment of these infections. A better identification and understanding of the factors that can affect transplacental transfer of maternal antibodies is crucial for optimization of vaccination strategies and close monitoring of particularly vulnerable newborns.

DETAILED DESCRIPTION:
The investigators aim to include 4050 patients and collect a maternal at delivery cord blood sample.

The aim of the investigators is to measure and compare ratio of transplacental transfer of maternal anti-virus antibodies according to the mode of acquisition of immunity (post-vaccination, or post-natural or mixed infection), gestational age at birth (< 32 Weeks of Gestation -WG-, 32-37 WG and > 37 WG) for several virus (Hepatitis B virus, Varicella zoster virus, Rubella virus, Measles, Influenza Virus, Mumps Virus, SARS-CoV-2, Cytomegalovirus, Herpes Simplex Virus 1 and 2, Respiratory Syncitial Virus, Parvovirus B19, HTLV). The investigators also aim to identify factors likely to influence negatively or positively transplacental transfer of maternal antibodies as maternal age, maternal ethnic origin, parity and gestation, sex of the newborn, maternal chronic or acute infection/disease occurring during pregnancy; Birth weight, vaccine boost carried out during pregnancy (etc.) will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years old ;
* Pregnant patient (single or multiple pregnancy) ;
* Gestational age at the time of inclusion > 22 Weeks of Gestation ;
* Patient affiliated or entitled to a french social security scheme ;
* Patient who expressed a non-objection to participate in the study.

Exclusion Criteria:

* Misunderstanding of the French language;
* Participation in another interventional trial of category 1. Participation in category 2 research, with minimal risks and constraints, will be left to the discretion of the investigator;
* Patient under curatorship or guardianship ;
* Patient's refusal to participate in the research.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women followed in the Gynecology-Obstetrics department for their pregnancy and/or at the time of their delivery
Sampling Method: Non-Probability Sample
Enrollment: 4050 (Estimated)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Measure the transplacental transfer ratio of maternal anti-virus antibodies according to the mode of acquisition of immunity, gestational age at birth of specific viruses | 15 months
  This is a descriptive study that aim to measure the ratio of transplacental transfer of maternal anti-virus antibodies according to the mode of acquisition of immunity (post-vaccination, or post-natural or mixed infection), gestational age at birth (< 32 WA, 32-37 WA and > 37 WA) for the following virus : Hepatitis B virus, Varicella zoster virus, Rubella virus, Measles, Influenza Virus, Mumps Virus, SARS-CoV-2, Cytomegalovirus, Herpes Simplex Virus 1 and 2, Respiratory Syncitial Virus, Parvovirus B19, HTLV.
  Ratios will be expressed in absolute values : "antibody level in the newborn (units/ml) / antibody level in the mother (units/ml).

SECONDARY OUTCOMES:
Compare transplacental transmission ratios of the different specific antibodies. | 15 months
  Ratios will be expressed in absolute values : "antibody level in the newborn (units/ml) / antibody level in the mother (units/ml)
Identify factors likely to influence transplacental transfer of the maternal antibodies as maternal age, ethnic origin, parity and gestation, sex of the child, maternal chronic or acute infection/disease occurring during pregnancy | 15 months
  Identify factors likely to influence negatively or positively transplacental transfer of the maternal antibodies as maternal age, maternal ethnic origin, parity and gestation, sex of the newborn, maternal chronic or acute infection/disease occurring during pregnancy,birth weight, vaccine boost carried out during pregnancy.
  Ratios will be expressed in absolute values : "antibody level in the newborn (units/ml) / antibody level in the mother (units/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Christelle VAULOUP FELLOUS, Doctor, Principal Investigator — Paul Brousse Hospital

IPD SHARING:
Plan to Share IPD: No